CLINICAL TRIAL: NCT01551966
Title: Evaluation of Wireless Capsule Endoscopy for the Detection and the Control of the Esophageal Varices in Children
Brief Title: Esophageal Capsule Endoscopy in Children
Acronym: PREVOCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010.644/48
Record Dates: First submitted 2012-03-08; First posted 2012-03-13 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2013-07

CONDITIONS: Portal Hypertension; Cirrhosis
Keywords: Esophageal varices; Portal hypertension in children; Wireless capsule endoscopy
MeSH Terms: conditions — Hypertension, Portal; Fibrosis; Esophageal and Gastric Varices | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- video capsule endoscopy (Experimental)
  Interventions: Device: Wireless esophageal capsule endoscopy ( PillCam Eso2)

INTERVENTIONS:
Device: Wireless esophageal capsule endoscopy ( PillCam Eso2) — This is a simple blind (blind for the lecture of the capsule endoscopy record) study to evaluate the diagnostic value of the capsule endoscopy for the detection and the control of esophageal varices, the feasibility, tolerance and safety of the capsule endoscopy compared to the conventional EGD under general sedation in children presenting with portal hypertension.
  During one week, the patients will undergo two exams (capsule endoscopy and EGD under general sedation). The exams will be done by two different physicians.
  For to asses the tolerance, after they completed both exams, the patients will be asked to answer a "comfort score" questionnaire.
  In order to asses the safety of the capsule endoscopy, the patients will be followed for adverse events during 3 weeks after the completion of the capsule endoscopy.
  Other Names: PillCam Eso2

SUMMARY:
The portal hypertension (PHT) is the main complication in patients presenting with cirrhosis. It can be the direct cause of bleeding by rupture of the esophageal or gastric varices and can also contribute to the development of ascites, hepatic encephalopathy and pleuropulmonary complications.

In the paediatric population presenting with the PHT, one of every two children develops varices and thus has a significant risk of bleeding. Safe and easy to use, the video capsule endoscopy (VCE) is now routinely used in children for the exploration of the small bowel. But the role of the VCE for examination of the other parts of digestive tract still needs to be evaluated.

For the esophagus, the VCE could allow the diagnosis without the need of general sedation. Recent studies have shown a good sensitivity and tolerance of this technique for the initial diagnosis of esophageal varices (EV) in adult patients presenting with portal hypertension, but it has not yet been validated for this indication.

The investigators hypothesize that the VCE could be used in children with similar results in term of efficacy, as for adults.

This prospective simple blind multicentre study (blind for the lecture of the capsule endoscopy record), will investigate the diagnostic value of the VCE compared to the conventional esophagogastroduodenoscopy (EGD) under general sedation for the detection and the control of esophageal varices in children.

If it is provided that the VCE is as efficient as it is for the adults, it could become a very interesting alternative to the conventional EGD because less expensive and less invasive. Moreover, this technique would be very useful as a means of early detection on the EV and/or their control.

ELIGIBILITY:
Inclusion Criteria:

* patients between 7 and 18 years old
* presenting a portal hypertension and/or cirrhosis
* patients who are referred for a conventional EGD under general sedation
* patients who are not participating in other clinical studies
* written informed consent obtained from the patient and his/her legal guardians.

Exclusion Criteria:

* patients presenting a contra indication for upper endoscopy or for the ingestion of the video capsule, especially those with clinical or radiological suspicion of upper gastrointestinal strictures (esophageal surgery or eosinophile esophagitys)
* patients presenting with dysphagia or gastrointestinal tract strictures (patients with Crohn's disease, small bowel carcinoma, stenosis due to the chronic use of a NSAI medication, acute necrotizing enterocolitis or prior abdominal surgery of the gastrointestinal tract); swallowing disorders with or without impaired consciousness;
* patients under calcium channel blocking agents medication;
* patient presenting with diverticulosis (Marphan's or Ehlers Danlos's syndrome)
* patients with cardiac pacemaker or other implanted electro medical device
* patients scheduled for a magnetic resonance imaging (MRI) examination within 7 days after ingestion of the capsule (and until the capsule is evacuated)
* any other life-threatening conditions.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic value of the wireless capsule endoscopy | 1 week
  The diagnostic value of the wireless capsule endoscopy as measured by the sensitivity of the wireless capsule endoscopy for the detection and the control of esophageal varices in children compared to the EGD sensitivity.

SECONDARY OUTCOMES:
Diagnostic value comparing the specificity, the positive and negative predictive value (PPV, NPV) of the wireless capsule endoscopy | 1 week
  Diagnostic value comparing the specificity, the positive and negative predictive value (PPV, NPV) of the wireless capsule endoscopy with the results for the EGD under general sedation.
Feasibility and safety of the wireless capsule endoscopy | 4 weeks
  Feasibility and safety of the wireless capsule endoscopy compared to the conventional EGD under general sedation as expressed by the safe completion of the wireless capsule endoscopy.
Acceptance of the wireless capsule endoscopy | 1 week
  Acceptance of the wireless capsule endoscopy by the patient compared to the EGD under general sedation by calculating a comfort score.
Applicability of the wireless capsule endoscopy | 1 week
  Applicability of the wireless capsule endoscopy by evaluating the ability to detect the esophageal or fundic varices, the presence of a portal hypertension gastropathy and the classification of the esophageal varices compared to the EGD results.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Service de Pédiatrie Médicale, Hôpital Pellegrin, CHU de Bordeaux, Bordeaux
  - Service d'Hépatologie, gastroentérologie et nutrition pédiatrique, Hôpital Femme Mère Enfant, Hospices Civils de Lyon, Bron
  - Clinique de Pédiatrie, Hôpital Jeanne de Flandre, CHU de Lille, Lille
  - Service de Gastroentérologie, Mucoviscidose et Nutrition, Hôpital Robert Debré, AP-HP, Paris
  - Service de Hépato Gastroentérologie et Nutrition, Hôpital Necker Enfants Malades, AP-HP, Paris
  - Service de Pédiatrie, Hôpital Sud, CHU de Rennes, Rennes
  - Service de Gastroentérologie, Hépatologie, Nutrition et Diabétologie, Hôpital des Enfants, CHU de Toulouse, Toulouse

REFERENCES:
- [Result] Cardey J, Le Gall C, Michaud L, Dabadie A, Talbotec C, Bellaiche M, Lamireau T, Mas E, Bridoux-Henno L, Viala J, Restier-Miron L, Lachaux A. Screening of esophageal varices in children using esophageal capsule endoscopy: a multicenter prospective study. Endoscopy. 2019 Jan;51(1):10-17. doi: 10.1055/a-0647-1709. Epub 2018 Sep 5. PMID 30184608